The COV-EAT: Dietary and Lifestyle Habits of Children and Adolescents and Their Parents During the Pandemic of COVID-19 in Greece.

**NCT Number: Not available yet** 

**Document Date: 03/06/2020** 

## **Study Protocol**

The aim of the COV-EAT study was to examine potential changes in children' and adolescents' dietary and lifestyle (physical activity, sedentary behavior and sleep) habits during the quarantine that was implemented in Greece due to COVID-19.

The COV-EAT study was a cross-sectional study, based on data collected at the end of lockdown period due to COVID-19 pandemic, in Greece. Specifically, the data were collected between 30/04/2020 and 24/05/2020.

An online survey was conducted in a random sample of families. Parents self-reported their child's and their own dietary and lifestyle habits, as well as information about their sociodemographic status. The questionnaire was self-reported by volunteers (parents of children aged 2-18 years). After extensive information about the aim of the study and their rights, the volunteers were requested to consent for their participation.

The survey consisted of 70 questions in 3 sections.

The first section focused on participants' sociodemographic data and included 15 questions, about gender, age, number of kids, city of residence and socioe-conomic level.

The second section contained 20 questions about parents' dietary and lifestyle habits before and during quarantine. Specifically, parents had to answer questions about the frequency of cooking at home and their fast-food consumption, the number of meals and snacks consuming per day, the reasons of snacking and their body weight and height.

The third section contained 35 questions about their child's eating habits and its sedentary behaviors. Parents had to answer about their child's body weight and height, the number of meals and snacks during the day, the frequency of breakfast, fast-food, fruits, juices, vegetables, dairy, red meat, poultry, fish, starch, legumes, sweets, salty snacks and beverages consumption, the servings of fruits, juices, vegetables and dairy consumed per day, the possible vitamin supplementation as well as screen time, sleep duration and changes in physical activity. All answers were given both before and during quarantine situation.

## Statistical Analysis Plan (SAP)

Descriptive statistics will be presented as means and SDs for continuous variables and frequencies and percentages for categorical variables. We will use paired t-tests to evaluate the significance of changes from pre-quarantine to quarantine in the responses. All statistical analyses will be performed using the statistical software package IBM SPSS statistics, version 23 (IBM Corporation). Significant differences or relations will be accepted at a p-value less than 0,05.

## **Informed Consent Form**

Dear Parents,

In this questionnaire, you are invited to take part voluntarily. The aim of the study is to investigate the potential changes in yours dietary and lifestyle habits as well as your children' during the quarantine due to the COVID-19 pandemic. The questionnaire is ANONYMOUS and it takes about 15 minutes to complete it. To participate in the study you must be a parent or guardian of a child aged 2-18 years.

If you agree with the personal data protection policy of this study, please select the corresponding field below by providing your consent.

Thank you in advance for your participation!

| $\square$ I declare that the data of this questionnaire are confidential and are $u$ | sed |
|---|---|
| anonymously for statistical analysis and scientific publication. | |
| □ I do not wish to participate in this study. | |